CLINICAL TRIAL: NCT02618447
Title: 4D Phase Contrast MR: Validation and Evaluation of Hypertrophy in Liver Cancer
Brief Title: 4D Phase Contrast MR: Hypertrophy in Liver Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 201406079
Record Dates: First submitted 2015-11-18; First posted 2015-12-01 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Liver Cancer; Cancer of the Liver
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Arm 1: 4D phase contrast MR scan (Experimental): * Each patient will undergo a total of 3 MRI/MRA scans (lasting 30-60 minutes):
    * Scan 1: Baseline (pre-portal vein embolization (PRE))
    * Scan 2: Early after PVE (within 48 hours)
    * Scan 3: Late after PVE (at 3-8 weeks).
  * Scans 1 and 3: routine liver MR sequences with/without contrast (Gadoxetic acid, Eovist) and 4D phase contrast of the portal venous system. The 4D phase contrast sequence will be repeated twice at each time point, adding about 15-30 minutes to each scan.
  * Scan 2: 4D phase contrast sequences and imaging for localization.
  Interventions: Device: 4Dimensional Phase Contrast Magnetic Resonance Angiography; Procedure: Portal vein embolization

INTERVENTIONS:
Device: 4Dimensional Phase Contrast Magnetic Resonance Angiography — 4D PC MRA is a new non-contrast MRA technique that can measure flow of blood within vessels of interest over time.
  Other Names: 4D PC MRA
Procedure: Portal vein embolization
  Other Names: PRE

SUMMARY:
The investigators hypothesize that 4Dimensional Phase Contrast Magnetic Resonance Angiography (4D PC MRA) evaluation of portal venous flow predicts underlying liver function and hypertrophic potential in patients with liver cancer presenting for portal vein embolization (PVE). 4D PC MRA may provide a non-invasive measure of liver function that could help determine which patients could safely and successfully undergo PVE and subsequent resection of tumor. By comparing 4D PC MRA results with invasive catheter measurements the investigators will validate the flow findings. Further regression/correlation analysis with functional measures of the liver (HIDA scans), volumetrics, Doppler flow analysis, histology, and outcomes will help the investigators to determine the ability of 4D PC MRA to predict functional status and hypertrophic potential of the liver prior to PVE and hepatectomy allowing for better patient selection and reduced morbidity/mortality.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of malignant liver tumor
* Clinically referred for portal vein embolization
* At least 18 years of age
* Willing and able to provide informed consent

Exclusion Criteria:

* Documented or reported contrast allergy
* Unable to receive or tolerate MRI scan after evaluation of MRI screening form
* GFR (glomerular filtration rate) < 30 on labs drawn within 6 weeks of imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-08-05 (Actual); Primary Completion 2016-02-04 (Actual); Study Completion 2016-02-04 (Actual)

PRIMARY OUTCOMES:
Ability of the 4D PC MRA to measure portal venous flow findings compared to reference standards of catheter-based flow quantification | Up to 6-8 weeks post PVE
  -Data from the 4D PC MRA will be compared with the reference standards of the catheter-based flow quantification to validate venous flow findings
Ability of the 4D PC MRA to measure flow velocities as compared to reference standards of the Doppler Flow Analysis | Up to 6-8 weeks post PVE
  -Data from the 4D PC MRA will be compared with the reference standards of the Doppler Flow Analysis to measure flow velocities
Ability of the 4D PC MRA to measure liver function | Up to 6-8 weeks post PVE
  -4D PC MRA results will be compared with invasive catheter measurements to validate the portal venous flow findings. Regression/correlation analysis will be used to analyze association between 4D PC MRA and liver function. Residuals will be tested for normality with the Shapiro-Wilk W test, and if residuals are non-normally distributed, the Spearman's rank correlation coefficient will be used
Ability of the 4D PC MRA to measure hypertrophic potential (liver function is preserved) | Up to 6-8 weeks post PVE
  -Data from the 4D PC MRA will be compared with the reference standards of the HIDA scan and biopsy specimens.
Ability of the 4D PC MRA to measure flow direction of flow as compared to reference standards of the Doppler Flow Analysis | Up to 6-8 weeks post PVE
  -Data from the 4D PC MRA will be compared with the reference standards of the Doppler Flow Analysis to measure direction of flow

CONTACTS AND LOCATIONS:
Overall Officials: Nael E Saad, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu